CLINICAL TRIAL: NCT04640298
Title: A Prospective Study of a Single Injection Cross-linked Sodium Hyaluronate Combined With Triamcinolone Hexacetonide (CINGAL®) to Provide Symptomatic Relief of Osteoarthritis of Hip Joint
Brief Title: Study of Cingal® for Symptomatic Relief of Osteoarthritis of Hip Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cingal 20-01
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Hip
Keywords: Sodium Hyaluronate; Triamcinolone Hexacetonide
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: CINGAL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cingal (Experimental): Single injection of Cingal into the hip joint of subjects diagnosed with osteoarthritis of the hip.
  Interventions: Device: Cingal

INTERVENTIONS:
Device: Cingal — Single injection into the hip joint of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH).

SUMMARY:
This Trial will obtain clinical data to support an expanded indication for a single injection of Cingal used for the symptomatic relief of osteoarthritis in the hip joint.

DETAILED DESCRIPTION:
Single injection into the hip joint of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH). Participants to be followed to 6 Months post-injection.

ELIGIBILITY:
Screening Inclusion Criteria:

1. Age 18 years or older
2. Body Mass Index (BMI) ≤ 35 kg/m2
3. Diagnosis of symptomatic osteoarthritic joint in the index hip (Kellgren-Lawrence grade I to III) to be treated with CINGAL injection.
4. Failed conservative treatment for joint osteoarthritis.
5. NRS on walking ≥4 and ≤ 9 in index hip.
6. Subject must be willing to abstain from other treatments of the index hip for the duration of the study.
7. Subject is willing to discontinue all analgesics including NSAIDs, except acetaminophen/paracetamol, at least seven days before the treatment injection and through the completion of the study.
8. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least forty-eight hours prior to the Baseline Visit and each follow-up assessment, the subject is willing to discontinue use of acetaminophen/paracetamol.
9. Subject is willing to maintain a stable dose of oral glucosamine and/or chondroitin sulfate products throughout the study, if taken prior to signing the informed consent form (ICF).
10. Able and willing to provide signed informed consent.

Baseline Inclusion Criteria

1. NRS pain on walking ≥4 and ≤ 9 in index hip

Screening Exclusion Criteria:

1. History of hypersensitivity to any of the ingredients in the hyaluronan or corticosteroids
2. Infection or skin disease in the area of the injection site or hip joint
3. NRS pain on walking > 3 the contralateral hip.
4. NRS pain on walking > 3 in the ipsilateral knee or ankle joints.
5. Subject received an injection of Hyaluronic Acid (HA) and/or steroid in either joint within 6 months of signing the informed consent form (ICF). A subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either joint during the course of this study.
6. Known inflammatory or autoimmune disorders (including rheumatoid arthritis, gout), or other pre-existing medical conditions that, in the opinion of the investigator, could impact treatment of the hip joint or affect the ability of the subject to accurately complete the study questionnaires and comply with the study requirements.
7. Subject is taking medications at the time of signing the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
8. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index hip only) corticosteroid within 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index hip is allowed.
9. Significant trauma to the index hip within 26 weeks of screening
10. Chronic use of narcotics or cannabis.
11. Ligament instability or tear in index hip.
12. Diagnosis of fibromyalgia
13. Diagnosis of osteonecrosis in index hip
14. Subject has significant varus or valgus deformity greater than 10 degrees in either knee.
15. Subject requires consistent use of an assistive device (e.g. wheelchair, walker, etc.) Occasional use of a cane is acceptable.
16. Uncontrolled diabetes with HbA1c of >7%.
17. Subject is a woman who is pregnant or breastfeeding at the Screening Visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
18. Subject is receiving or in litigation for worker's compensation.
19. Otherwise determined by the investigator to be medically unsuitable for participation in this study.

Baseline Exclusion Criteria

1. Subject has a decrease of ≥ 2 in the NRS pain on walking from Screening to Baseline in the index hip.
2. Subject has a contraindication to continue with the study treatment injection based on the visual appearance of the synovial fluid aspirate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Mezger, Study Director — Anika Therapeutics
Locations (4):
- Krajská zdravotní, a.s. - Masarykova nemocnice Ústí nad Labem, o.z., Ústí nad Labem, Czechia
- Poland (3):
  - NZOZ MEDI-SPATZ M.Spatz, Gliwice
  - SPORTO sp. z o.o, Lodz
  - Przychodnia Rodzinna na Sadowej, Torun

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cingal
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT)
Arm/Group | Cingal
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Index Hip [Count of Participants; unit: Participants]
  Right | 17
  Left | 8

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain on Walking
Description: Reduction of Index Hip Numerical Rating Scale (NRS) Pain on Walking from baseline to 6 months post injection was obtained from participant responses. The NRS Pain Score is an 11-point Likert scale ranged from 0 = No Pain to 10 = Worst Pain Level. A negative value for the change in NRS Pain Score indicates less pain post-treatment. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: 6 months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cingal: Single injection of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH)
Arm/Group | Cingal
Number analyzed (Participants) | 25
score on a scale | -2.48 (1.61)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

2. Secondary Outcome: Lequesne Hip Index
Description: Improvement from baseline to 6 months in The Lequesne Hip Index. The Lequesne Hip Index is a three-section patient questionnaire that evaluates (1) pain or discomfort, (2) maximum distance walked, and (3) activities of daily living with 0 = best results / normal scores, to scores >14 = extremely severe, to a maximum index score of 24 points.
  A negative value for the change in Lequesne Hip Index indicates improvement. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
score on a scale | -2.76 (2.57)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

3. Secondary Outcome: Patient Global Assessment (PGA) Score
Description: The change from baseline to 6 months in hip pain post-treatment as measured by the Patient Global Assessment (PGA) Score. PGA Score records participant responses to their assessment of how much their STUDY (treated) hip is bothering them today . The PGA Score is a validated 11-point Likert scale ranged from 0 = No Pain to 10 = Worst Pain.
  A negative value for the change from baseline indicates improvement in PGA Score. A larger negative value indicates less pain, and a better clinical outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
score on a scale | -2.56 (1.73)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

4. Secondary Outcome: The Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. A Calculated Percentage (%) of Participants Responding to Treatment
Description: The post-treatment responder rate is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder to treatment. The criteria for response are (1) improvement in pain or physical function >50% and an absolute change >20 mm; or (2) improvement of >20% with an absolute change >10 mm in at least of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cingal
Number analyzed (Participants) | 25
Participants | 18

5. Secondary Outcome: Usage of Rescue Medication (Acetaminophen/Paracetamol). Number of Participants NOT Using Rescue Medication.
Description: The usage of Rescue Medication (RM) as based on the number of participants at 6 Months post treatment that were NOT using acetominophen/paracetamol RM for pain or discomfort.
  A larger percentage of participants that were NOT using RM may correlate to a better clinical outcome in terms of pain.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cingal
Number analyzed (Participants) | 25
Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the time of the baseline study visit until study completion at 6 Months.
Description: The definitions of adverse event (AE) and serious adverse event (SAE) are the same as used in the clinicaltrials.gov definitions.
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE) were collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | Cingal
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 4/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=25)
Headache (Nervous system disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats associated with the conduct of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INVESTIGATOR may publish the Data/Results with the consent of the SPONSOR if:

1. Publication is done after primary publication covering data from all participating sites, and provided the Data/Results do not contain any Confidential Information.
2. Eighteen (18) months has elapsed after entire completion of the Clinical Trial at all participating sites.

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT04640298/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04640298/SAP_001.pdf